CLINICAL TRIAL: NCT03027401
Title: Clinical Sequencing of Cancer and Tissue Repository: ClinOmics
Brief Title: Clinical Sequencing of Cancer and Tissue Repository: OncoGenomics
Status: Withdrawn | Type: Observational
Why Stopped: closed by PI and FDA
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 170040; 17-C-0040
Record Dates: First submitted 2017-01-19; First posted 2017-01-23 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Neoplasms; Adenomatous Polyposis Coli; Neurofibroma, Plexiform; Myelodysplastic Syndromes
Keywords: Genetic Testing; Tumor Profiling; Biorepository
MeSH Terms: conditions — Neoplasms; Adenomatous Polyposis Coli; Neurofibroma, Plexiform; Myelodysplastic Syndromes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group A: Adult/pediatric with suspected or confirmed malignancy, family history of malignancy, undergoing surgery with no malignancy; tissues collected previously under CLIA or for research.

SUMMARY:
Background:

Saliva, blood, tissue, and cancer contain DNA. DNA makes the "instruction book" for the cells in the body. Cancer is caused by changes in DNA that affect cell function. Researchers want to test DNA of people with tumors. They want to look for genetic changes in tumors that could be targets for treatment. Because DNA can change as cancer changes, more testing may be done at different times.

Objectives:

To find the DNA changes in cancer that may help guide treatment. To collect samples and data to be used in future studies.

Eligibility:

People any age with cancer or a pre-cancerous tumor

Design:

* Participants will be screened with a medical history, physical exam, and blood tests. Participants will give a sample of their tumor. This is usually from a previous procedure. Participants will give a saliva or blood sample. They cannot eat, drink, smoke, or chew gum for 30 minutes before giving saliva. They will spit about 1 teaspoon of saliva into a tube.
* Some participants may have a punch biopsy instead. A small instrument will take a small piece of skin.
* Researchers will collect data from participants medical records.
* Participants will answer questions about their family health history. They will also answer questions about their views on the study, including possible unexpected results.
* Extra blood or tissue samples may be taken at other times during the participants' treatment. All samples will be saved in secure ClinOmics freezers to be used in future studies.
* Participants will be told by their doctors if any test results affect their health or their cancer treatment.

DETAILED DESCRIPTION:
Background:

* Laboratory-based investigations have contributed to an improved understanding of the biology of cancer and to the development of new therapies for malignancies.
* Omics investigation may identify novel drivers in the germline or tumor for high risk, relapsed, refractory or rare cancers.
* Omics investigation may identify germline or somatic alterations that are medically actionable and or can enable precision therapy.

Objectives - Primary Objective:

-Identify incidental and secondary findings in germline DNA and actionable somatic mutations for reporting clinical results from a CLIA-certified lab into CRIS medical records.

Eligibility - Adult or Pediatric patients of any age with one of the following:

* Diagnosis of any tumor, malignancy, pre-malignant disorder, or suspected cancer susceptibility familial syndromes, regardless of patient age; OR
* Individuals without history of malignancy who are undergoing surgery; OR
* Individuals without a history of cancer but evidence of an inherited cancer syndrome based on family history and/or other manifestations of a pre-cancerous syndrome (e.g. polyposis, plexiform neurofibromas, myelodysplastic disease); OR
* Patient enrolled in an approved companion protocol.
* Tissue (including tumor, normal, blood, bone marrow, serum, plasma, or other tissues) that has been previously collected under CLIA and maintained in a CLIA lab which is available for CLIA analysis.
* Tissue (including tumor, normal, blood, bone marrow, serum, plasma, or other tissues) that has been previously collected and is available for research analysis.
* Biospecimens can be collected with minimal additional risk to the subject during sampling or procedures required for routine patient care.
* Individual may be undergoing treatment for malignancy, premalignant condition or receiving other care associated with an inherited cancer syndrome.
* Patients may be referred to the Principal Investigator from outside institutions.
* Ability of subject or Legally Authorized Representative (LAR) to understand and the willingness to sign a written informed consent OR
* IRB waiver of the requirement for informed consent for specific types of tissue.

Design:

* This study will allow for the collection of specimens for CLIA reporting of germline and somatic mutations. The study will also collect specimens for a Tissue Repository, and for other investigations as outlined below.
* CLIA testing activities will include

  * DNA extracted from a section of tumor, malignant tissue, blood, or bone marrow samples for somatic mutation sequence analysis
  * Germline DNA extracted from lymphocytes, saliva, skin, or any normal uninvolved tissues for sequence analysis to identify somatic alterations in the cancer and for the reporting of incidental findings of established clinical validity and utility.
* Research activities may include:

  * DNA, RNA and protein Omics analyses from extracted normal and/or tumor tissues; the remainder of the tumor tissue will be stored.
  * Germline DNA and RNA analyses from extracted lymphocytes or other normal uninvolved tissue.
  * T (TCR) or B Cell Receptor sequencing from blood, tumor, or malignant tissue.
  * Establishing Patient-Derived Models such as patient-derived xenografts (PDXs), early-passage in vitro tumor cultures, and organoid cultures, conditionally reprogrammed cells (CRC) lines, explant and cell lines from tumor or normal samples by the NCI Patient-Derived Models Repository (PDMR) at Frederick National Laboratory for Cancer Research or by the OncoGenomics laboratory.
  * Cryopreservation of viable normal (e.g. PBMC) or malignant tissues.
  * Establishment of EBV transformed cell lines from blood for medical research either by Coriell Institute or by investigators on this protocol.
  * Omics (Genomics, Proteomic, Epigenetics, Metabolomics) studies will be performed.
* Expected accrual 50-500 patients per year. Total protocol accrual goal 5,000 patients.

ELIGIBILITY:
* INCLUSION CRITERIA:

Adult or Pediatric patients with one of the following:

* Diagnosis of any tumor, malignancy, pre-malignant disorder, or suspected cancer susceptibility familial syndromes, regardless of patient age; OR
* Individuals without history of malignancy who are undergoing surgery; OR
* Individuals without a history of cancer but evidence of an inherited cancer syndrome based on family history and/or other manifestations of the syndrome (i.e. polyposis, plexiform neurofibromas, myelodysplastic syndrome); OR
* Tissue (including tumor, normal, blood, serum, plasma, or other tissues) that has been previously collected under CLIA and maintained in a CLIA lab which is available for CLIA analysis.
* Tissue (including tumor, normal, blood, bone marrow, serum, plasma, or other tissues) that has been previously collected and is available for research analysis.
* Biospecimens can be collected with minimal additional risk to the subject during sampling or procedures required for routine patient care.
* Individual may be undergoing treatment for malignancy, premalignant condition or receiving other care associated with an inherited cancer syndrome.
* Ability of subject or Legally Authorized Representative (LAR) to understand and the willingness to sign a written informed consent; OR
* IRB waiver of the requirement for informed consent for specific types of tissue.

EXCLUSION CRITERIA:

-None

Max Age: 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Samples for the population cohort will be selected from patients that are co-enrolled on other NIH protocols (both inpatient and outpatient) as well as community referrals from outside NIH.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-01-10 (Actual); Primary Completion 2020-10-05 (Actual); Study Completion 2020-10-05 (Actual)

PRIMARY OUTCOMES:
Identify incidental and secondary findings in germline DNA and actionable somatic mutations for reporting clinical results from a CLIA-certified lab into CRIS medical records. | ongoing
  Sample analysis.

SECONDARY OUTCOMES:
Molecular, genomic, epigenetic, transcriptomic, proteomic, metabolomics and other "omics" profiling on tumors, malignancies and normal tissues | ongoing
  Sample analysis for identification of biomarkers, drivers and medically actionable targets for clinical management.
Create a tissue repository | ongoing
  Repository for analysis of samples.
Extraction and storage of circulating tumor DNA | ongoing
  Storage of samples.
Establishing Patient-derived models | ongoing
  Analysis of samples.
Cryopreservation of viable tumor tissue for future study | ongoing
  Sample storage for future analysis.
Establishment of EBV transformed cell lines for research | ongoing
  Analysis of germline samples.
Creation of an OncoGenomics oversight committee | ongoing
  Oversight and development of new treatment approaches.
Assessment of effects of the informed consent process | ongoing
  Survey data collection and analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Javed Khan, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Green RC, Berg JS, Grody WW, Kalia SS, Korf BR, Martin CL, McGuire AL, Nussbaum RL, O'Daniel JM, Ormond KE, Rehm HL, Watson MS, Williams MS, Biesecker LG; American College of Medical Genetics and Genomics. ACMG recommendations for reporting of incidental findings in clinical exome and genome sequencing. Genet Med. 2013 Jul;15(7):565-74. doi: 10.1038/gim.2013.73. Epub 2013 Jun 20. PMID 23788249
- [Background] Weiner C. Anticipate and communicate: Ethical management of incidental and secondary findings in the clinical, research, and direct-to-consumer contexts (December 2013 report of the Presidential Commission for the Study of Bioethical Issues). Am J Epidemiol. 2014 Sep 15;180(6):562-4. doi: 10.1093/aje/kwu217. Epub 2014 Aug 22. PMID 25150271
- [Background] Appelbaum PS, Waldman CR, Fyer A, Klitzman R, Parens E, Martinez J, Price WN 2nd, Chung WK. Informed consent for return of incidental findings in genomic research. Genet Med. 2014 May;16(5):367-73. doi: 10.1038/gim.2013.145. Epub 2013 Oct 24. PMID 24158054
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2017-C-0040.html